CLINICAL TRIAL: NCT06824623
Title: Multicenter Prospective Observational Study to Prevent the Risk of REadmission and DEhydration of Patients With ileoSTOmy in Elective Colorectal Surgery
Brief Title: Readmission and Dehydration Prevention in Patients With Elective Ileostomy
Acronym: PREDESTO
Status: Recruiting | Type: Observational
Sponsor: Multidisciplinary Italian Study group for STOmas (MISSTO) (Other)
Collaborators: Convatec Limited (Unknown)
Responsible Party: Sponsor
Other Study IDs: MISSTO-02
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Ileostomy - Stoma; Colorectal Surgery; Dehydration
Keywords: ileostomy; colorectal cancer; inflammatory bowel disease; dehydration; readmission; colorectal surgery
MeSH Terms: conditions — Dehydration; Colorectal Neoplasms; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ileostomy patients: Consecutive patients undergoing ileostomy creation after elective colorectal resection

SUMMARY:
The goal of this prospective observational study is to evaluate the adherence to DRIP score calculation and the application rate of each proposed item to prevent dehydration and readmission in patients undergoing ileostomy creation after elective colorectal resection different Italian colorectal surgical centers.

The primary endpoint is to verifythe application rate of DRIP score calculation and protocol items.

Secondary endpoints are 30, 90, and 180-day total and dehydration readmission rates.

DETAILED DESCRIPTION:
Introduction Ileostomy is often performed for patients with conditions such as inflammatory bowel disease or colorectal cancer. However it introduces unique challenges for postoperative care, including the risk of dehydration and hospital readmission. Dehydration is a common complication in patients with ileostomies, due to the loss of fluids and electrolytes through the stoma output. Unlike normal bowel function, the output from an ileostomy is more liquid and can lead to significant fluid depletion if not carefully managed. This risk is exacerbated in the immediate postoperative period when patients adjust to their altered physiology. Failure to maintain adequate hydration and electrolyte balance can result in severe complications, including acute kidney injury and metabolic imbalances, necessitating readmission to the hospital. Readmission rates among patients with ileostomies remain a significant concern in healthcare, contributing to increased healthcare costs and patient burden. Studies indicate that dehydration accounts for a substantial proportion of these readmissions, underscoring the need for effective strategies to manage and prevent this complication. Patient education, tailored hydration plans, and close monitoring are critical components of care to mitigate this risk. Understanding the interplay between ileostomy function, dehydration, and readmissions is essential to improve outcomes for these patients. The Dehydration Readmission After Ileostomy Prediction (DRIP) scoring system is a novel, validated scoring system of patient and clinical factors that can be used to identify patients at risk of being readmitted for dehydration after ileostomy creation.

The DRIP protocol The DRIP score has been proposed by Chen et al. in 2018 and it includes some items, considered as risk factors for readmission after ileostomy creation. In table 1 there is a complete description of DRIP score calculation and items. The suggested interventions have been proposed to reduce the risk of dehydration and readmission: pre-discharge ostomy education; discharge home with intravenous fluids infusion; discharge home with antidiarrheal drugs; daily home nursing follow-up; daily phone follow-up; outpatient postoperative follow-up within seven days (with blood tests). Based on DRIP score calculation, patients are classified into 5 categories: very low, low, medium, high and very high risk.

Study design:

This is a multicenter, prospective observational study, to evaluate the application rate of DRIP score and the application rate of different strategies of care for ileostomy patients in different Italian colorectal surgical centers.

The following parameters will be evaluated for all patients: in-hospital stoma care, post-op i.v. rehydration, post-operative creatinine, outpatient follow-up after discharge, pre-discharge ostomy education. The DRIP score will be calculated for each patient.

Additional parameters will be evaluated for patients at medium, high and very high-risk of dehydration (based on DRIP score classification): discharge home with intravenous fluids infusion; discharge home with antidiarrheal and/or absorbent drugs; discharge home with specific alimentary regimen; home care with nursing follow-up; daily phone follow-up; postoperative clinic follow-up within 14 days with laboratory tests.

Methods:

Data will be prospectively collected from 01/05/2025 to 30/04/2026, with 6-months follow-up from 01/05/2026 to 30/09/2026.

Each participating center will decide how best to identify eligible patients. Data will be entered directly onto the secure electronic REDCap database by study collaborators at the participating hospital sites using pseudonymised data.

The following data will be considered:

Age Operation date (ileostomy creation) Preoperative stoma-nurse counselling Preoperative stoma siting Sex ASA BMI Clinical frailty index Chronic Kidney Disease Preoperative creatinine value Hypertension Diabetes Indication for surgery (rectal cancer, colon cancer, IBD, diverticulitis, other) Operative approach: open, laparoscopic, robotic ERAS protocol Operation type (Rectal or colon resection, total colectomy, IPAA, SB resection, other) Previous or associated small bowel resection Distal ileostomy (<30cm from ileocecal valve) Stoma siting respect Pre-discharge ostomy education Post-operative i.v. rehydration (day of interruption) Post-op worst creatinine value Ileostomy output at discharge: quality (bristol scale grade) and quantity (cc) Discharge date Postoperative early (<30d) complications (based on Clavien-Dindo classification) Postoperative late (>30d) complications (based on Clavien-Dindo classification) Postoperative early (<30d) stoma complications Postoperative late (>30d) stoma complications Readmission Date of readmission Cause of readmission (dehydratation, renal failure, other complication) Discharge home with intravenous fluid rehydration Discharge home with antidiarrheal medication Home care nursing follow-up (at least 3 times a week) Phone follow-up (at least 3 times a week) Post-discharge clinic follow-up within 14 days with laboratory tests Ileostomy closure date

Sample size calculation:

Based on previous experience of the steering committee of the study during the study period we expect to collect approximately 300 patients. Assuming a 20% readmission rate this number will provide the possibility to collect about 50 patients with readmission in order to evaluate risk factors for readmission.

Statistical analysis Statistical analysis will be performed using Chi-square or Fisher's exact probability tests for categorical variables or Student's t test for continuous variables. Multivariable logistic regression analysis will be used to identify predictors of readmission. A p-value <0.05 will be considered statistically significant. Statistically significant factors associated with readmission and dehydration in the univariate analysis, as well as clinically relevant factors regardless of statistical significance, will be included in the model.

ELIGIBILITY:
Inclusion Criteria:

* All patients with elective ileostomy performed during the study period for benign or malignant colorectal disease
* Age > 18 years
* Written consent

Exclusion Criteria:

* Emergency surgery
* Other ostomy than ileostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing ileostomy creation after elective colorectal resection in different Italian colorectal surgical centers.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
DRIP score calculation and protocol items | From enrollment to the end of recruitment at 6 months
  Application rate of DRIP score calculation and protocol items

SECONDARY OUTCOMES:
Readmission rates | From enrollment to the end of recruitment at 6 months
  30, 90, and 180-day total and dehydration readmission rates

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Ferrara, MD, Principal Investigator — Multidisciplinary Italian Study group for STOmas (MISSTO)
Locations (7):
- Italy (7):
  - ASST Ovest Milanese, Ospedale di Legnano, Legnano, Italy
  - Luigi Sacco University Hospital, Milan, Italy
  - Università degli Studi Milano-Bicocca, Ospedale San Gerardo, Monza, Italy
  - University of Palermo, "Paolo Giaccone" University Hospital, Palermo, Italy
  - Ospedale Santa Maria della Misericordia, Rovigo, Italy
  - ASST Nord Milano, Ospedale Città di Sesto San Giovanni, Sesto San Giovanni, Italy
  - IRCCS Policlinico di Bologna, Bologna

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferrara F, Parini D, Bondurri A, Veltri M, Barbierato M, Pata F, Cattaneo F, Tafuri A, Forni C, Roveron G, Rizzo G; Multidisciplinary Italian Study group for STOmas (MISSTO). Italian guidelines for the surgical management of enteral stomas in adults. Tech Coloproctol. 2019 Nov;23(11):1037-1056. doi: 10.1007/s10151-019-02099-3. Epub 2019 Oct 12. PMID 31606801
- [Background] Parini D, Bondurri A, Ferrara F, Rizzo G, Pata F, Veltri M, Forni C, Coccolini F, Biffl WL, Sartelli M, Kluger Y, Ansaloni L, Moore E, Catena F, Danelli P; Multidisciplinary Italian Study group for STOmas (MISSTO). Surgical management of ostomy complications: a MISSTO-WSES mapping review. World J Emerg Surg. 2023 Oct 10;18(1):48. doi: 10.1186/s13017-023-00516-5. PMID 37817218
- [Background] Ferrara F, Rizzo G, Bondurri A, Forni C, Anania G, Anastasi A, Baiocchi GL, Boccia L, Cassini D, Catarci M, Cestaro G, Cillara N, Cobellis F, De Luca R, De Nardi P, Deidda S, Delogu D, Fedi M, Giuffrida MC, Grossi U, Impellizzeri H, Langone A, Lauretta A, Lo Celso F, Maffioli A, Manigrasso M, Marafante C, Marano L, Marinello P, Massucco P, Merlini D, Morelli L, Mozzon M, Pafundi DP, Pata F, Pellino G, Peltrini R, Petrina A, Piazza D, Rabuini C, Resendiz A, Salmaso B, Santarelli M, Sena G, Siragusa L, Tamini N, Tondolo V, Tutino R, Vannelli A, Veltri M, Vincenti L, Parini D; MISSTO Snapshot Study Collaborative Group. Outcomes of loop ileostomy after rectal resection for cancer: A prospective observational multicenter snapshot study from Multidisciplinary Italian Study group for STOmas (MISSTO). Tech Coloproctol. 2024 Dec 11;29(1):16. doi: 10.1007/s10151-024-03047-6. PMID 39661237
- [Background] Chen SY, Stem M, Cerullo M, Canner JK, Gearhart SL, Safar B, Fang SH, Efron JE. Predicting the Risk of Readmission From Dehydration After Ileostomy Formation: The Dehydration Readmission After Ileostomy Prediction Score. Dis Colon Rectum. 2018 Dec;61(12):1410-1417. doi: 10.1097/DCR.0000000000001217. PMID 30303886